CLINICAL TRIAL: NCT01169857
Title: Velcade for Proliferative Lupus Nephritis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants were enrolled.
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X05321; 1003010960 (Other: Weill Cornell Medical College IRB)
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Lupus Nephritis; Proteinuria; Hematuria
Keywords: Proliferative lupus nephritis; WHO class III/IV/V lupus nephritis; Proteinuria; Hematuria; Velcade; SLE; Bortezomib; Proteasome inhibitor
MeSH Terms: conditions — Lupus Nephritis; Proteinuria; Hematuria | interventions — Bortezomib; Proteasome Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Velcade Therapy (Experimental)
  Interventions: Drug: Velcade

INTERVENTIONS:
Drug: Velcade — Velcade at 1.3 mg/m2, on days 1, 4, 8 and 11 (=1 cycle). The study will involve 3 cycles of Velcade therapy.
  Other Names: Bortezomib; Proteasome inhibitor

SUMMARY:
The primary objective is to test the safety and efficacy of Velcade to induce remission in WHO class III/IV/V lupus nephritis that are refractory to standard medications.

DETAILED DESCRIPTION:
This exploratory single center, open-label, single treatment group assignment, safety, and efficacy study will enroll 14 patients with WHO class III/IV/V lupus nephritis. Subjects will receive 12 doses of Velcade to induce clinical remission.

ELIGIBILITY:
Inclusion Criteria:

1. ACR criteria for lupus (minimum 4 out of 11).
2. Biopsy proven WHO class III or IV or V lupus nephritis with clinical activity.
3. GFR must be greater or equal to 30 cc/min/1.73 m2.
4. Proteinuria must exceed 1000 mg per day except for WHO class V lupus nephritis, daily proteinuria must be greater or equal to 2000 mg.
5. Primary therapy for active disease must have been given at least 6 months prior to protocol enrollment for WHO lupus III/IV.

Exclusion Criteria:

1. Serum creatinine of more than 3.0 mg/dL on repeated testing.
2. Greater than 50% fibrosis on renal biopsy.
3. Platelet count of less than 30× 109/L.
4. Absolute neutrophil count of less than 1.0 × 109/L.
5. Greater than or equal to Grade 1 peripheral neuropathy.
6. Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure.
7. Hypersensitivity to Velcade, boron or mannitol.
8. Serious medical conditions and infections (including HIV, HCV, HBV) or psychiatric illness.
9. Known history of untreated positive PPD.
10. Serious complications from systemic lupus such as cerebral lupus and severe active infections.
11. Diagnosed or treated for another malignancy within 3 years of enrollment.
12. Greater than 1.5x upper limit of normal total bilirubin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Proteinuria | 1 year
  Quantification of 24 hr urinary protein.

SECONDARY OUTCOMES:
Renal function | 1 year
  Serum creatinine and GFR
Lupus activity score | 1 year
  Assessment of SELENA-SLEDAI

CONTACTS AND LOCATIONS:
Overall Officials: Choli Hartono, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States